CLINICAL TRIAL: NCT06058832
Title: Effects of Low-intensity Shockwave Therapy Versus Kegel Exercises on Arteriogenic Erectile Dysfunction in Diabetic Patients
Brief Title: Effects of Low-intensity Shockwave Therapy Versus Kegel Exercises on Arteriogenic Erectile Dysfunction in DM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elsayed Hassan Elsayed Abosteit, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shockwave in ED
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Sexual Dysfunction; Shock Wave
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-intensity Shockwave Therapy (Experimental): patients will receive 6 sessions, once per week of low-intensity extracorporeal shock wave with the following parameters: - 3000 SWs (energy intensity of 0.09 mJ/mm2) to each of five different sites: three along the penile shaft and two at the crural level plus Sildenafil 25mg of daily dose and 50mg on-demand dose one hour before intercourse for 6 weeks.
  Interventions: Device: Low-intensity Shockwave Therapy
- Kegel Exercises (Experimental): kegel exercises plus sildenafil 25mg of daily dose and 50mg on-demand dose one hour before intercourse for 6 weeks.
  Interventions: Other: Kegel Exercises
- control group (No Intervention)

INTERVENTIONS:
Device: Low-intensity Shockwave Therapy — patients will receive 6 sessions, once per week of low-intensity extracorporeal shock wave with the following parameters: - 3000 SWs (energy intensity of 0.09 mJ/mm2) to each of five different sites: three along the penile shaft and two at the crural level plus Sildenafil 25mg of daily dose and 50mg on-demand dose one hour before intercourse for 6 weeks.
  Arms: Low-intensity Shockwave Therapy
Other: Kegel Exercises — * The patient was asked to perform short (1 second) and long-lasting (6-10 seconds) contractions of the target muscles. Later, the exercises will do with the patient sitting or standing.
  * Patient asked to repeat the contractions daily. Each patient performed 15 short and 15 long-lasting contractions in a prone, sitting, or standing position. Patients asked to do 30 contractions in the morning 30 contractions in the evening
  Arms: Kegel Exercises

SUMMARY:
* To assess the effectiveness of low-intensity shockwave therapy (Li-ESWT) in the management of Arteriogenic erectile dysfunction in diabetic patients.
* To assess the effectiveness of Kegel Exercises in the management of Arteriogenic erectile dysfunction in diabetic patients.
* To compare the effectiveness of Li-ESWT and Kegel Exercises in the management of Arteriogenic erectile dysfunction in diabetic patients.

DETAILED DESCRIPTION:
Erectile dysfunction is defined as the persistent inability to attain and maintain an erection enough to permit satisfactory sexual performance. Although ED is a benign disorder, it may affect physical and psychosocial health and may have a significant impact on the quality of life of sufferers and their partners.

According to the underlying causes, ED can be classified as psychogenic, endocrinologic, neurogenic, and vasculogenic. Vasculogenic erectile dysfunction is defined as an inability to get or keep an erection firm enough for sexual intercourse due to diseases such as diabetes mellitus and atherosclerotic vascular occlusive disease .

ED has been reported to occur in ≥50% of men with DM worldwide. It is usually present within 10 years of diagnosis of DM. The incidence of ED was reported to be higher in men with DM than for men without DM and up to 12% of men who present with ED were found to have previously undiagnosed DM.

Low-intensity extracorporeal shock wave therapy (Li-ESWT) was used in both in vitro and in vivo studies and the results showed that this energy can stimulate angiogenesis. The idea of applying Li-ESWT to the penis came from animal studies in which Li-ESWT was applied to the myocardium of pigs, where it has been reported that there was an improvement in ischemia-induced myocardial dysfunction.

Low-intensity extracorporeal SW therapy (Li-ESWT) of the penis would improve penile blood flow and endothelial function by stimulating angiogenesis in the corpora.

Oral phosphodiesterase-5 inhibitors (PDE-5 inhibitors), such as sildenafil and tadalafil, are usually the first-line treatment of erectile dysfunction. They are effective in a wide range of etiologies including cardiovascular disease, diabetes, and hypogonadism.

Contraction of the ischiocavernosus participates in the process of enhancing erectile rigidity by compressing the roots of the corpora cavernosa and inducing short-term suprasystolic intracavernosal pressures.

Further, bulbospongiosus contraction leads to temporary engorgement of the glans penis and corpus spongiosum and results in similar short-term increases in intra spongiosal pressures.

ELIGIBILITY:
Inclusion Criteria:

1. Ninety married men were diagnosed with T2DM participated in this study.
2. The patients complained from arteriogenic ED > 6 months (Reisman et al., 2015) before the participation in this study
3. All patients aged between 35-55 years old.
4. Glycated hemoglobin (HbA1c) less than 9%.
5. Body mass index of the patients was < 30 Kg/m2.

Exclusion Criteria:

1. Alcohol-abuse, illegal drug consumer patients.
2. Patients with cardiac diseases that prevent or affect sexual activity (heart attack, stroke, heart failure, myocardial infarction life-threatening, arrhythmia, etc within the previous 6 months).
3. Patients with any pulmonary, liver, or kidney diseases.
4. Patients with neurological insults, spinal cord injuries, stroke, polyneuropathy, etc.
5. Patients with diagnosed psychiatric/mental complaints.
6. Patients with blood pressure of more than 140/90 mmHg.
7. Patients with peripheral vascular disease.
8. Patients with venogenic ED.
9. Patients with past radical prostatectomy, extensive pelvic surgery, or previous pelvic trauma.
10. Patients recovering from cancer in the past 5 years
11. Penile anatomical abnormalities.
12. Patients with clinically significant chronic hematological disease.
13. Patients who received Anti-androgens or radiotherapy treatment of pelvic region.
14. Patients with untreated hypogonadism.
15. Patients with psychogenic ED (normal nocturnal penile tumescence parameters)
16. Patient with penile prosthesis

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Penile color-coded Duplex scanning | baseline
  for exclusion of psychogenic and venogenic erectile dysfunction (ED) and confirm arteriogenic ED. It will be used at baseline and post-intervention.
International Index of Erectile Function (IIEF-EF) questionnaire | baseline
  At baseline and post-intervention, patients will be assessed and scored according to the five-item version of the International Index of Erectile Function (IIEF-5), which consists of five questions. Its score ranges from 1 to 25 and classifies ED severity with the following breakpoints: severe (1-7/25), moderate (8-11/25), mild to moderate (12-16/25), mild (17-21/25), and no ED (22-25/25)

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed Abosteit, PhD, Principal Investigator — physical therapy
Locations (1):
- Alhussein Hospital, Cairo, Egypt

REFERENCES:
- [Background] Cohen D, Gonzalez J, Goldstein I. The Role of Pelvic Floor Muscles in Male Sexual Dysfunction and Pelvic Pain. Sex Med Rev. 2016 Jan;4(1):53-62. doi: 10.1016/j.sxmr.2015.10.001. Epub 2016 Jan 8. PMID 27872005
- [Background] Dorey G, Speakman M, Feneley R, Swinkels A, Dunn C, Ewings P. Randomised controlled trial of pelvic floor muscle exercises and manometric biofeedback for erectile dysfunction. Br J Gen Pract. 2004 Nov;54(508):819-25. PMID 15527607
- [Background] Gruenwald I, Kitrey ND, Appel B, Vardi Y. Low-Intensity Extracorporeal Shock Wave Therapy in Vascular Disease and Erectile Dysfunction: Theory and Outcomes. Sex Med Rev. 2013 Jul;1(2):83-90. doi: 10.1002/smrj.9. Epub 2015 Oct 18. PMID 27784587